CLINICAL TRIAL: NCT00956332
Title: Phase I/IIa Safety, Two-dose Study of MultiGeneAngio in Patients With Chronic Critical Limb Ischemia
Brief Title: Safety Study of MultiGeneAngio in Patients With Chronic Critical Limb Ischemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MultiGene Vascular Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGVS-MGA 002
Record Dates: First submitted 2009-08-09; First posted 2009-08-11 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease; Critical Limb Ischemia
Keywords: Peripheral arterial disease (PAD); Peripheral vascular disease (PVD); Critical limb ischemia (CLI); Cell therapy; Gene therapy; Endothelial cells; Smooth muscle cells; Angiogenesis; Arteriogenesis; amputation; diabetic foot
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGA - Low therapeutic dose (Experimental)
  Interventions: Biological: MultiGeneAngio
- MGA - Intermediate therapeutic dose (Experimental)
  Interventions: Biological: MultiGeneAngio

INTERVENTIONS:
Biological: MultiGeneAngio — Low-therapeutic dose of MultiGeneAngio in suspension administered as one treatment, intra-arterially
  Arms: MGA - Low therapeutic dose
Biological: MultiGeneAngio — Intermediate-therapeutic dose of MultiGeneAngio in suspension administered as one treatment, intra-arterially
  Arms: MGA - Intermediate therapeutic dose

SUMMARY:
The purpose of this study is to evaluate the safety and activity of two doses of MultiGeneAngio, a cell therapy product produced from the patient's own cells, as potential treatment for patients with chronic critical limb ischemia.

DETAILED DESCRIPTION:
Approximately 16 million patients worldwide (1 in 20 people over the age of 50) suffer from peripheral arterial disease(PAD). PAD is characterized by narrowing or occlusion of vessels supplying blood to the lower limbs, most often due to atherosclerosis. Symptoms of PAD include claudication that may progress to critical limb ischemia manifested by rest pain, tissue loss and gangrene, which eventually may necessitate amputation.

MultiGeneAngio is a cell therapy-based product developed for treatment of patients with chronic critical limb ischemia due to narrow or blocked leg arteries. MultiGeneAngio is composed of endothelial and smooth muscle cells that are isolated from a short vein segment harvested from the patient's arm. After isolation the cells are expanded, characterized, and gene modified by transfer of angiogenic genes.

MultiGeneAngio is a clear cell suspension injected intra-arterially at the site of blockage using a standard diagnostic catheter, in order to create and expand new collateral arteries, and thereby improve blood flow to an ischemic limb.

Comprehensive pre-clinical studies, as well as clinical experience with PAD patients suffering from claudication showed that production and administration of MultiGeneAngio was feasible and safe, as no apparent drug-related adverse events have been observed. Moreover, follow-up data of peak walking times imply a beneficial trend of this efficacy end-point. Additional follow-up data will continue to be collected to help evaluate the safety and efficacy of MultiGeneAngio.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 50 years of age or older
* Ischemic rest pain (Rutherford category 4) and/or
* Non-healing wounds (Rutherford category 5)
* ABI of 0.5 or less, or TBI of 0.3 or less
* Ankle systolic pressure of 70 mm Hg or less, or toe systolic pressure of 50 mm Hg or less
* Poor or no option for conventional revascularization

Exclusion Criteria:

* Life expectancy of less than one year
* Presence of significant inflow disease (>50% stenosis) in the distal aorta, common or external iliac
* Advanced CLI, characterized by extensive tissue loss or gangrene (Rutherford category 6)
* Previous major amputation on the leg to be treated or planned major amputation within a month from enrollment
* Evidence of osteomyelitis
* Ischemic wounds with uncontrolled infectious symptoms
* Heart angioplasty or CABG within 3 months prior to enrollment
* Severe congestive heart failure (New York Heart Association stage IV)
* Acute cardiovascular event within 3 months prior to enrollment
* Uncontrolled blood pressure: SBP≥ 180 mmHg or DBP ≥110 mmHg
* Known Buerger's disease
* History of bleeding diathesis (e.g., hemophilia due to Factor VIII or IX deficiency)
* Renal failure defined as a serum creatinine >2.5mg/dL
* Significant hepatic disease:>3-fold elevation in ALT/AST, HBV or HCV carriers
* Severe pulmonary disease
* Active proliferative retinopathy and/or severe macular oedema
* Intra-ocular surgery within 6 months prior to enrollment
* Immunodeficient states (e.g. known HIV positivity, or organ transplant recipient) or subject receiving immunosuppressive medication
* History of malignant neoplasm (except curable non-melanoma skin malignancies) within 5 years prior to enrollment
* Pregnant or lactating women
* Previous treatment with angiogenic growth factors or stem cells
* No demonstrable venous access
* Known hypersensitivity to VEGF, Angiopoietin-1, or heparin

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The safety of MultiGeneAngio will be assessed by monitoring adverse events | Up to 15 years after treatment

SECONDARY OUTCOMES:
Improvement in critical limb ischemia symptoms | Up to 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sam L. Teichman, MD, Study Director — Independent consultant
Locations (7):
- Israel (7):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital, Ein Kerem, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Chaim Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Background] Staudacher DL, Preis M, Lewis BS, Grossman PM, Flugelman MY. Cellular and molecular therapeutic modalities for arterial obstructive syndromes. Pharmacol Ther. 2006 Jan;109(1-2):263-73. doi: 10.1016/j.pharmthera.2005.08.005. Epub 2005 Oct 21. PMID 16243400
- [Background] Gray BH, Conte MS, Dake MD, Jaff MR, Kandarpa K, Ramee SR, Rundback J, Waksman R; American Heart Association Writing Group 7. Atherosclerotic Peripheral Vascular Disease Symposium II: lower-extremity revascularization: state of the art. Circulation. 2008 Dec 16;118(25):2864-72. doi: 10.1161/CIRCULATIONAHA.108.191177. No abstract available. PMID 19106409
- [Background] Staudacher DL, Flugelman MY. Cell and gene therapies in cardiovascular disease with special focus on the no option patient. Curr Gene Ther. 2006 Dec;6(6):609-23. doi: 10.2174/156652306779010705. PMID 17168694
- [Background] Gluzman Z, Koren B, Preis M, Cohen T, Tsaba A, Cosset FL, Shofti R, Lewis BS, Virmani R, Flugelman MY. Endothelial cells are activated by angiopoeitin-1 gene transfer and produce coordinated sprouting in vitro and arteriogenesis in vivo. Biochem Biophys Res Commun. 2007 Jul 27;359(2):263-8. doi: 10.1016/j.bbrc.2007.05.097. Epub 2007 May 25. PMID 17544375
- [Background] Tongers J, Roncalli JG, Losordo DW. Therapeutic angiogenesis for critical limb ischemia: microvascular therapies coming of age. Circulation. 2008 Jul 1;118(1):9-16. doi: 10.1161/CIRCULATIONAHA.108.784371. No abstract available. PMID 18591450
- [Background] Isner JM, Vale PR, Symes JF, Losordo DW. Assessment of risks associated with cardiovascular gene therapy in human subjects. Circ Res. 2001 Aug 31;89(5):389-400. doi: 10.1161/hh1701.096259. PMID 11532899